CLINICAL TRIAL: NCT01837459
Title: Vascular Function in Children With Obstructive Sleep Apnea
Brief Title: A Research Study for Children About Heart Changes and Obstructive Sleep Apnea (OSA)
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CIN001VF; R01HL080670-01A2 (NIH)
Record Dates: First submitted 2013-04-08; First posted 2013-04-23 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Sleep Disordered Breathing; Vascular function; Arterial stiffness; Polysomnography; Cytokines
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Obese-Normal: Obese with Apnea Hypopnea index (AHI) <1
- Obese-SDB: Obese and with AHI>1
- Lean-Normal: Non-obese with AHI<1
- Lean-SDB: Non-obese with AHI>1

SUMMARY:
In this research study the investigators want to learn more about the risk of developing blood vessel and heart disease from night-time sleep apnea. Sleep apnea is a condition that results from blocking of the throat during sleep. This study examines changes in blood pressure, blood vessel stiffness, heart size and levels of specific substances in the blood which may cause heart disease.

This study is for children ages 5 to 13 years. The study involves 3 visits over 18 months. The first and last visits include an overnight sleep study (polysomnography or PSG). All the visits will include:

* body measurements to measure growth and how weight is distributed,
* resting blood pressure measurements,
* heart measurements (electrocardiogram and ultrasounds of the heart and blood vessels),
* 36 hour home ambulatory blood pressure measurements,
* blood tests to look at things like fats, cholesterol, inflammatory factors,
* questionnaires

Optional parts of the study include DNA and for children 8 years and older, testing and questionnaires to learn more about how sleep relates to learning, memory and behavior issues.

DETAILED DESCRIPTION:
This study is designed primarily to investigate the changes in blood vessels compliance and stiffness in children ages 5 to 13 years with the syndrome of obstructive breathing during sleep. It is designed to examine the relationship of the severity of the syndrome to vascular functions and to specific inflammatory mediators related to early stages of arterial stiffness and their effect on cardiovascular end-points, namely twenty-hour ambulatory blood pressure and left ventricular mass. The study will also examine the relationship between plasma and tonsillar tissue levels of inflammatory cytokines, and as well as the relationships between obstructive breathing during sleep and children's attention and problem-solving skills. Our aim is to identify vascular risk factors in childhood and to determine whether sleep disordered breathing in children represents an independent risk factor for cardiovascular disease and neurodevelopmental deficits which if left inadequately identified could track into adult years

* Hypothesis that increased levels of inflammatory cytokines will correlate with severity of the OSA disorder.
* Hypothesis that severity of the OSA disorder will correlate with measures of increased arterial wall stiffness, which in turn will lead to an increase in pulse pressure and left ventricular mass.

This study will examine the vascular function in children, both lean and obese, with the syndrome of obstructive breathing during sleep which encompasses children with varying degrees of sleep disordered breathing (SDB). Children included in the SDB groups will have OSA above 1 obstructive episode per hour of sleep. The standard of care for a child with symptoms of obstructive breathing during sleep in otolaryngology practices is to undergo a tonsillectomy and or adenoidectomy (T&A). Children with SDB and who are scheduled to have T&A will be followed for 18 months and compared to children without SDB. To discern the effect of obesity on vascular function from the effects of sleep disordered breathing (SDB), the study will consist of four groups. Two groups, one lean and one obese, will have SDB and two groups, one lean and one obese, will be normal controls. Efforts will be made to match subjects across all groups. There is the potential that all groups will not contain the same number due to differences in incidence of OSA in relation to weight.

There are 3 visits over approximately 18 months. The first visit will function as a qualifying visit based on the Obstructive Index from the polysomnography (OI>1 for SDB group and OI<1 with no snoring for the control group). Visits are approximately 9 months apart with the first and last visit including overnight polysomnography (PSG). Tonsillar tissue specimens will be obtained from a subset of SDB subjects who are scheduled for T&A.

Data captured will include:

* Blood will be measured for high-sensitivity C reactive protein (hsCRP), serum amyloid A, cytokine panel, fasting lipoprotein analysis, complete blood count (CBC), glucose, insulin direct renin and DNA (optional).
* Tonsillar tissue will be measured for hsCRP, serum amyloid A, cytokine panel.
* Anthropometrics including height, weight, arm and finger circumferences, neck circumference, waist to hip ratio, and arm lengths.
* Left ventricular structure and vascular stiffness measurements include echocardiogram, carotid ultrasound, and radial tonometry.
* Resting blood pressure measurements include a continuous beat to beat BP recording obtained by a Portapres monitor with ECG and respiration monitoring done throughout sleep during the PSG and 30 minutes while awake in the morning.
* Activity and home ambulatory blood pressure (AMBP)measurements will be continuously monitored (every 30 minutes) using an automated oscillometric BP monitor over a 36 hour period simultaneously with actigraphy.
* Questionnaires about sleep and QOL.
* A subset of subjects aged 8 and older can participate in a neurobehavioral component that includes a formal assessment of attention and problem-solving.

ELIGIBILITY:
Inclusion Criteria:

* Normal controls will be enrolled from children who have a signed informed consent and who have completed the initial polysomnography; whose history does not reveal any symptoms of obstructive breathing during sleep; and who have a polysomnogram that is considered normal.
* SDB groups will be enrolled from children who have a signed informed consent and who have completed the initial polysomnography with OI>1; whose history includes snoring, hypertrophied tonsils or hypertrophied adenoids. Subjects will be assigned to a study group based on results of the overnight polysomnogram.

Exclusion Criteria:

Exclusion criteria:

* Children with positive history of snoring without evidence of AHI> 1 and who do not follow through with tonsillectomy or adenoidectomy surgery.
* Children with chronic pulmonary conditions including asthma (children with mild, intermittent asthma will be included and are defined as use of rescue inhaler < 1/wk unless treatment for exercise induced asthma).
* Children with cardiac disease
* Children with neuromuscular disorders
* Children with developmental delay such as Down syndrome
* Children with chronic renal disease such as chronic pyelonephritis or glomerulonephritis
* Children with endocrinological disorders or who are on chronic steroid therapy including inhaled steroids.
* Children using medications which influence the autonomic nervous system such as adrenergic and cholinergic drugs, alpha and beta blockers, and drugs with parasympatholytic action.
* Children with any acute or chronic inflammatory condition.
* Children with BMI Z score that exceeds 2.9 for age and gender.
* Children who do not complete the first 36 hour AMBP study with a 70% success rate of BP readings.
* Children with a history of chronic or recurrent tonsillitis (by parent or physician report) defined as 6 episodes of tonsillitis / year for a period of one year; 5 episodes of tonsillitis / year for 2 years; 4 episodes of tonsillitis / year for 3 years.

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children 5-13 years recruited from the community, otolaryngology and sleep disorder clinics
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2006-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Comparison across groups of change in levels of C-reactive protein and cytokines | Baseline, 9 months, 18 months

SECONDARY OUTCOMES:
Comparison across groups of changes in carotid and aortic compliance and stiffness as measured in changes in pulse waves, and carotid intima media thickness (mm) | Baseline, 9 months, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Raouf Amin, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
Analysis is in progress and may take up to an additional year due to complexity of data.

REFERENCES:
- [Derived] Witter AM, Smith DF, Khan MTF, Nakamura A, Schuler CL, DiFrancesco MW, Hossain MM, Amin RS. Relationship of Circadian Blood Pressure Dysregulation With Left Ventricular Structure and Function in Children With Obstructive Sleep Apnea. J Sleep Res. 2025 Oct;34(5):e70049. doi: 10.1111/jsr.70049. Epub 2025 Apr 1. PMID 40170220
- [Derived] Domany KA, Huang G, Hossain MM, Schuler CL, Somers VK, Daniels SR, Amin R. Effect of Adenotonsillectomy on Cardiac Function in Children Age 5-13 Years With Obstructive Sleep Apnea. Am J Cardiol. 2021 Feb 15;141:120-126. doi: 10.1016/j.amjcard.2020.11.019. Epub 2020 Nov 19. PMID 33220319